CLINICAL TRIAL: NCT05671211
Title: Effects Of Task-Oriented Training on Balance,Walking,Functional Mobility,Activities Of Daily Living and Quality Of Life In Individuals With Stroke
Brief Title: Effects Of Task-Oriented Training In Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Ozkeskin, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOzkeskin747
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stroke; Tas-Oriented Training; Balance; Walking; Mobility; Activities of Daily Living; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in control group will receive an exercise program consisted of upper and lower extremity strengthening and balance exercises.The exercises will be started as 8-10 repetitions and one set and the number of sets will be increased according to the progression of the patient. Exercises will be applied for 6 weeks, 5 days a week, for a total of 30 sessions, each session for 1 hour.
  Interventions: Other: Conventional Therapy
- Task-Oriented Training Group (Experimental): Participants in the task-oriented training group will receive the same treatment given to the control group, with an additional 30 minutes of task-oriented training.Task-Oriented Training Program will include several everyday tasks (Getting up from the chair, walking 10 steps taking a book from the table and walking backwards to sit on the chair,Walking forward and sideways over obstacles...etc.).The exercises will be started as 12-15 repetitions and 1 set at the beginning, and the number of sets will be increased according to the progression of the patient. A total of 30 sessions will be applied, 5 days a week for 6 weeks, with a total of 1.5 hours of exercises.
  Interventions: Other: Task-Oriented Training

INTERVENTIONS:
Other: Task-Oriented Training — Participants in this group will receive 30 minutes of task-oriented training and 1 hour of conventional therapy for 6 weeks 5 times a week.
  Arms: Task-Oriented Training Group
Other: Conventional Therapy — Conventional therapy will be consisted of balance,upper and lower extremity strengthening exercises.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate the effects of task-oriented training on balance,functional mobility,walking, activities of daily living and quality of life in individuals with stroke.

DETAILED DESCRIPTION:
Eligible participants will be randomized to task-oriented group or control group.Control group will receive conventional therapy generally consisted of neurophysiological approaches for 6 weeks 5 times a week for 1 hour per session.Task-oriented group will receive conventional therapy and task-oriented training for 6 weeks 5 times a week 1,5 hours per session.Each participant will be assessed before and after the 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Modified Rankin score between 0-3
* Having a stroke for the first time
* At least 1 month has passed since the stroke
* Able to walk 10 M with or without assistance
* Having a Mini Mental Test score of 24 and above
* Volunteering to participate in the study
* Being fluent in Turkish language

Exclusion Criteria:

* Having an additional neurological disease other than stroke
* Having an additional disease that prevents mobility
* Having a condition that prevents you from exercising
* Receiving an existing additional medical treatment for spasticity treatment
* Having a history of multiple strokes
* Having severe visual problems post stoke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale(BBS) | six weeks
  BBS, evaluates daily activities including static sitting and standing balance, as well as transfers, turning, and picking up objects from the ground, in 14 items.Scoring is given as 0-4. It scores from 4 (normal performance) to 0 (not able to do the movement) according to the person's ability to do what is asked of them safely and independently. The total score is 56 points. 0-20 indicates high risk, 21-40 indicates medium risk, and 41-64 indicates low risk.
10 Meter Walking Test(10MWT) | siz weeks
  This test calculates the unassisted walking speed of individuals at a distance of 10 meters. In this test, the person will be asked to walk at their normal pace in a pre-measured 10 meter area.
Timed Up And Go Test (TUG) | siz weeks
  It is a frequently used test that evaluates functional mobility and dynamic balance. At the beginning of the test, individuals sit in a chair. A distance of 3 m is set in front of the patient. With the start command, the patient gets up from his seat and walks 3 m, turns around and walks back and sits. With the start command, the time until the moment of sitting on the chair is recorded in seconds.Shorter duration indicates better functional mobility.
Stroke-Specific Quality of Life Scale(SS-QOL) | six weeks
  The Stroke-Specific Quality of Life Scale evaluates the quality of life in post-stroke individuals.
  It consists of 49 items from 12 areas;energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision, work/productivity. Each item is evaluated on a 5-point Likert scale. Maximum score is 245, high scores indicates good quality of life.

SECONDARY OUTCOMES:
5 Times Sit to Stand Test(5XSST) | six weeks
  The 5 Repetitive Sit-Rise Test (5XSST) is a practical test that evaluates lower extremity functional strength and balance.The individual rests on a standard 43 cm chair, arms crossed over shoulders, feet on the floor.Individual will be asked to sit and stand up quickly 5 times. Duration of 5 repetitions will be recorded in seconds.Results below 15 seconds indicate good stability, while 15 seconds and above indicate impaired balance and function.
Functional Ambulation Classification (FAC) | six weeks
  Functional Ambulation Classification (FAC) is a common clinical gait assessment method. Walking ability is scored between 0-5 according to the amount of support needed during the training and classification is made over 6 categories.. 5 points indicate fully independent ambulation while 0 points indicate non-functional ambulation .
Functional Independence Scale (FIM) | six weeks
  Functional Independence Scale is used to evaluate activities of daily living.- It consists of a total of 18 items(13 physical,5 social) that include cognitive status assessment. Each item is scored between 1 and 7. 7 means that the specified item is performed completely independently, while 1 indicates the need of full assistance. The maximum score that can be obtained from the scale is 126, indicating good performance. The lowest score is 18 and shows poor performance.

CONTACTS AND LOCATIONS:
Overall Officials: ALI E. MUTLU, mD, Principal Investigator — Bornova Ozilhan State Hospital Physical Therapy unit
Locations (1):
- Bornova Türkan Ozilhan State Hospital Physical Therapy Unit, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No